CLINICAL TRIAL: NCT03774992
Title: Clinical Study Of Nearsightedness, TReatment With Orthokeratology Lenses 2
Acronym: CONTROL2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Collaborators: Ens Eyes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CONTROL2
Record Dates: First submitted 2018-12-11; First posted 2018-12-13 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Myopia
Keywords: Orthokeratology lenses; Myopia; Children
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orthokeratology (Experimental): Subjects randomized to OKL in the CONTROL-study
  Interventions: Device: Orthokeratology lenses
- Cross over (Experimental): Subjects randomized to SVS in the CONTROL-study
  Interventions: Device: Orthokeratology lenses

INTERVENTIONS:
Device: Orthokeratology lenses — Custom fit, form stable contact lenses

SUMMARY:
Myopia is a common disease of the eye with increasing prevalence all over the world including Denmark where the prevalence has increased from 12,8% in 2004 among young adults (mean age 19,3 years) till 17,9% in 2017 among school children (mean age 15,4 years). High myopia is associated with an increasing risk of sight threatening complications such as retinal detachment, glaucoma, macular choroidal degeneration, and myopic choroidal neovascularization. In myopia the eye is elongated compared to an emmetropic eye. If the elongation of the eye can be controlled the progression of myopia can be controlled. Asian studies have shown reduction in axial length growth by 36-46% in children using orthokeratology contact lenses (OKL). OKL are custom fit, form stable lenses. During sleep the cornea is reshaped creating an emmetropic vision during the day, so no glasses or contact lenses are needed.

In the CONTROL-study 60 Danish children aged six to 13 years were randomized 1:1 to either OKL (intervention group) or single vision spectacles (SVS) (control group) and followed for 18 months to compare changes in axial length (AL). In CONTROL2 the intervention group will be followed for another 18 month and the control group will be crossed over to OKL treatment.

The aims of CONTROL2 is to:

1. Investigate changes in axial length after 3 years of OKL wear (DreamliteR, Procornea, Nederlands).
2. Investigate changes in progression rate 18 month before and after OKL wear.
3. Investigate correlations between changes in choroidal thickness and changes in AL.
4. Investigate the safety of OKL treatment (Efron score).
5. Investigate changes in quality of life before and after OKL treatment using Pediatric Refractive Error Profile 2 (PREP2).
6. Investigate correlations between AC/A-ratio, peripheral refraction and higher order aberrations on myopia progression.

DETAILED DESCRIPTION:
Myopia is a common disease of the eye with increasing prevalence in the Western World as well as in South East Asia where 60-90% of the children are affected. A Danish study found that early debut of myopia is associated with a higher degree of myopia later on in life. Myopia may be corrected with spectacles, contact lenses or surgically, but despite this socio-economic burden, high myopia is associated with an increasing risk of sight threatening complications such as retinal detachment, glaucoma, macular choroidal degeneration and myopic choroidal neovascularization.

Myopia is a complex disease with a multi-factorial etiology. Twin studies and family studies have shown a high heritability for development of myopia, and more than 40 genetic loci have been identified. Outdoor activity seems to reduce the myopia progression. The shape of the eye may be of importance; axial growth makes the eye ellipsoidal which increase the peripheral defocus on the retina. Peripheral defocus has been suggested to induce further axial growth of the eyeball.

Accommodation is a significant covariant of near work and reading. A cross section study has shown a reduced precision in accommodation (A) on a near object combined with increased convergence (C) in myopic eyes. This increased AC/A ratio (dynamic) may be a predictor for myopia progression.

Interventions for reducing myopia progression have been many. The effects of progressive additional lenses, multifocal lenses and bifocal lenses have been limited. Anticholinergic eyedrops (Atropin 0.01%) significantly reduce the progression of myopia in Asian children by approximately 50% over a period of two years with limited side effects. Almost similar results have been found in Asian children using orthokeratology contact lenses (OKL) for reducing myopia progression.

OKL are custom fit, form stable lenses used during sleep. The lenses induce a temporary flattening of the cornea, which modify or eliminate refractive errors, leaving no need for glasses or contact lenses during daytime. OKL were introduced in the 1960 ́s, but with limited success due to lens material (PMMA) which was not gas-permeable. Decentration was also a problem making the effect variable and unpredictable. With new gas permeable lens materials and computer assisted topographic measurements of the cornea, fitting of the lenses has been improved significantly, so that nightly wear is now standard treatment.

A clear-cut reduction in axial length growth in Asian children using OKL compared to single-vision spectacles (SVS) has been proofed in several studies. In these studies, which are very heterogeneous regarding design, reductions of 36-46% in axial length growth were found compared to a matched control group. Two European prospective cohort studies have investigated the effect of OKL compared to SVS in Spanish children. A reduction in axial growth of 32 % and 38% respectively was found. Side effects of OKL have been evaluated; in a meta-analysis from 2015, including 8 Asian and one of the European studies. Odds Ratio for side effects were 8.87 for the OK group compared to the control group, however all side effects were mild and disappeared after termination of the treatment.

Thus, a reduction in childhood myopia using OKL has been proofed in Asian children; however, weather similar result can be achieved in a group of children from Northern Europe is unknown and to address that the CONTROL-study was conducted. The CONTROL-study is an eighteen-months randomized prospective 1:1 study of the progression of myopia in a group of Danish children wearing OKL nightly (n=30) compared to a control group wearing SVS (n=30). The study is ongoing and thus there are not yet published any results. However, the study has formed the basis for a unique opportunity to

1. Look at the long-term effects of OKL treatment (3 years) in regards to efficacy and safety, and
2. Evaluate the progression-rate of myopia 18 months prior to treatment compared to 18 months after treatment with OKL.

Primary goals of the CONTROL2:

1. To investigate changes in axial length after 3 years of OKL wear (DreamliteR, Procornea, Nederlands).

2. To investigate changes in progression rate 18 month before and after OKL wear.

1. To investigate correlations between changes in choroidal thickness and changes in AL.
2. To investigate the safety of OKL treatment (Efron score).
3. To investigate changes in quality of life before and after OKL treatment using Pediatric Refractive Error Profile 2 (PREP2).
4. To investigate correlations between AC/A-ratio, peripheral refraction and higher order aberrations on myopia progression.

ELIGIBILITY:
Inclusion Criteria:

* subjects enrolled in the CONTROL-study

Exclusion Criteria:

* none

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Axial length | 18 months
  Change in axial length (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Flemming Møller, Dr. med, Principal Investigator — Vejle Hospital and University of Southern Denmark
Locations (1):
- Vejle Hospital, Vejle, Jylland, Denmark